CLINICAL TRIAL: NCT02864160
Title: Integrated Second Language Learning for Chronic Care: A Model to Improve Primary Care for Hispanics With Diabetes
Brief Title: Integrated Second Language Learning for Chronic Care
Acronym: ISLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Arizona (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60045178; R01DK104648 (NIH)
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus
Keywords: Language Concordance; Diabetes Self-Management; Health Coaching; Latinos
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 2 group study with concurrrent random assignment to intervention or control group using random assignment list that was pre-generated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental): The health coaching intervention group (n=100) will receive written educational materials on diabetes self-management in Spanish and the diabetes self-management tools (stretch band, a glucometer, and a diabetes cookbook in Spanish). In addition, patients in the intervention group will be assigned a health coach who will provide health coaching over the course of 6 months with 14 phone calls.
  Interventions: Behavioral: Health Coaching
- Comparison group (Active Comparator): The comparison group (n=100) will receive the standard diabetes care that is offered at Heart of Ohio clinics including consultations with a primary care provider, a dietician, a pharmacist, and a diabetes educator. The comparison group will receive written educational materials on diabetes self-management in Spanish and diabetes self-management tools including a stretch band, a glucometer, and a diabetes cookbook in Spanish.
  Interventions: Behavioral: Comparison Group

INTERVENTIONS:
Behavioral: Health Coaching — Life style coaching in 3 in-person meetings and 14 phone calls; written educational materials; self-management tools (stretch band, a glucometer, and a diabetes cookbook in Spanish).
  Arms: Health Coaching
Behavioral: Comparison Group — Written educational materials; self-management tools (stretch band, a glucometer, and a diabetes cookbook in Spanish).
  Arms: Comparison group

SUMMARY:
Language barriers continue to impede access to quality care for limited English proficient populations. Recent research has demonstrated that access to language concordant providers increases quality of care. This project evaluates the efficacy and acceptability of a model intervention to improve second language proficiency, patient-centered communication, and clinical competency of nurse practitioner students who care for Spanish-speaking patients with diabetes.

DETAILED DESCRIPTION:
The purpose of this randomized controlled 2-group study is to test the effect of an innovative educational intervention called Integrated Language Learning for Chronic Care (IL2L) on successful self-management of diabetes. It pursues an integrated development of second language and interpersonal communication skills that will facilitate productive interactions between Spanish-speaking nurse practitioners (NP) and limited English proficiency Hispanic patients with diabetes. The intervention targets the acquisition of language skills that facilitate communicative functions known to be effective in engaging chronically ill patients. It accelerates acquisition of these skills by adding a longitudinal clinical instruction dimension. Further, the investigators propose that the efficacy of the intervention can be demonstrated at the provider level through improved linguistic and interpersonal performance and at the patient level through improved diabetes outcomes in response to language concordance. In support of these claims, the investigators seek to achieve the following specific aims:

Aim 1: To determine the efficacy of the IL2L for Chronic Care intervention on physical and mental health outcomes for Spanish-speaking patients with diabetes. Our hypothesis is: H1: Patients in the IL2L care group will report better physical health (HbA1C, lipids, and weight), mental health (depression and anxiety) and satisfaction with their healthcare than patients in the non-IL2L care group.

Aim 2: To determine the efficacy of the IL2L for Chronic Care intervention on provider language proficiency and interpersonal communication skills. Our hypothesis is:H2: Providers exposed to the IL2L intervention will demonstrate improved Spanish language skills and interpersonal communication skills upon completion of the intervention.Specific Aim 3: To assess the acceptability of the IL2L for Chronic Care model within a graduate level nurse practitioner curriculum in a leading College of Nursing.

The study will employ a mixed-methods model to assess the efficacy and accessibility of the IL2L for Chronic Care educational intervention in The Ohio State University's College of Nursing nurse practitioner program. To achieve Aim 1, the investigators will use a randomized control trial to demonstrate efficacy of the IL2L for Chronic Care model at the patient level. The investigators will compare a group of patients exposed to providers who underwent the IL2L intervention (intervention group) and a group of patients who are undergoing standard care (comparison group). To achieve Aim 2, the investigators will use a qualitative data interaction analysis system to demonstrate improvement in Spanish language proficiency and interpersonal communication skills. To achieve Aim 3, the investigators will use a combination of quantitative and qualitative measures within the RE-AIM model to assess the acceptability of the IL2L for chronic care model at the program level in a nurse practitioner program in a leading College of Nursing. The study has been approved by the institutional review boards of both universities prior to implementation and patients and student providers provide written informed consent.

ELIGIBILITY:
INCLUSION CRITERIA

Students:

Enrolled in nurse practitioner programs at Ohio State University or University of Arizona Minimum intermediate Spanish language fluency by Oral Proficiency testing Patients Self identify as Hispanic/Latino Self identify preference for health care interaction in Spanish Clinical diagnosis of Type 2 diabetes Hemoglobin A1C of 7 or higher 22 years or older Must have access to land line or mobile phone

EXCLUSION CRITERIA

Students:

Distinguished Spanish language fluency by Oral Proficiency testing Received professional training for a health-related profession in a Spanish-speaking country

Patients:

Clinic diagnosis of diabetic retinopathy, diabetic neuropathy, or diabetic nephropathy Clinical diagnosis of major depression Clinical diagnosis of other psychiatric disorder

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in Patient Hemoglobin A1C from Baseline to 6 Months | From baseline to 6 months
  Hemoglobin A1C is measured via a blood test and measures the patient's average plasma glucose concentration over the past 3 months and is reported as a percentage. In general, normal A1C levels for people without diabetes is 4% to 5.6% while a level of 5.7% of 6.4% indicates prediabetes, and 6.5% or above indicates diabetes.

SECONDARY OUTCOMES:
Change in Patient Self-Efficacy from Baseline to 6 Months as Assessed by the DSES | From baseline to 6 months
  Numerical score measured by the Diabetes Self-Efficacy Scale (DSES) which measures self-perceptions held by people with diabetes about their personal competence, power, and resourcefulness for successfully managing their diabetes. The scale has eight 10-point Likert-type items with lower scores indicative of higher self-efficacy, as defined by Grossman et al. (1987).
  Grossman HY, Brink S, Hauser ST. Self-efficacy in adolescent girls and boys with insulin-dependent diabetes mellitus. Diabetes care 1987;10(3):324-9.
Change in Patient Depression from Baseline to 6 Months as Assessed by the PHQ-9 | From baseline to 6 months
  Numerical score measured by the Patient Health Question-9 questionnaire which measures depression severity with Likert-type items ranging from 0 (not at all) to 4 (everyday), with higher scores indicative of greater depression. A score between 10 and 14 indicates moderate depression as defined by Spitzer et al. (2000).
  Spitzer RL, Williams JB, Kroenke K, Hornyak R, McMurray J. Validity and utility of the PRIME-MD patient health questionnaire in assessment of 3000 obstetric- gynecologic patients: the PRIME-MD Patient Health Questionnaire Obstetrics- Gynecology Study. Am J Obstet Gynecol 2000;183(3):759-69.
Change in Patient Anxiety from Baseline to 6 Months as Assessed by the GAD-7 | From baseline to 6 months
  Numerical score measured by the Generalized Anxiety Disorder questionnaire, a 7-item, 4-point Likert-type scale ranging from (0) Not at all to (3) Every day, with higher scores indicating greater functional impairment related to the patient's experience of anxiety. A score of greater than or equal to 10 indicates moderate anxiety, as defined by Spitzer et al. (2006).
  Spitzer RL, Kroenke K, Williams JBW, Löwe B. A Brief Measure for Assessing Generalized Anxiety Disorder: The GAD-7. Arch Intern Med. 2006;166(10):1092-1097.
Change in Patient Blood Pressure from Baseline to 6 Months | From baseline to 6 months
  Measured in mmHG. Normal blood pressure for most adults is defined as a systolic pressure of less than 120 and a diastolic pressure of less than 80. Elevated blood pressure is defined as a systolic pressure between 120 and 129 with a diastolic pressure of less than 80.
Change in Patient Weight from Baseline to 6 Months | From baseline to 6 months
  Measured in pounds and ounces
Change in Patient Body Mass Index from Baseline to 6 Months | From baseline to 6 months
  Measured in weight (kg)/height (m^2). In general, a Body Mass Index (BMI) of under 18.5 falls within the underweight range, 18.5 to 24.9 falls within the normal or Healthy Weight range, 25.0 to 29.9 falls within the overweight range, and 30.0 or higher falls within the obese range.
Change in Patient Waist Circumference from Baseline to 6 Months | From baseline to 6 months
  Measured in inches.
Change in Patient Total Cholesterol from Baseline to 6 Months | From baseline to 6 months
  Milligrams per deciliter of blood (mg/dL) that is reported as a whole number. In general, less than 200 mg/dL is considered normal, 200 to 239 mg/dL is borderline high, and at or above 240 mg/dL is high.
Change in Health Coach Spanish Language Proficiency from Baseline to 6 Months as Assessed by the ACTFL | From baseline to 6 months
  Standardized Oral Proficiency score American Council on the Teaching of Foreign Languages (ACTFL) 2012 proficiency scale. Levels range from Distinguished (highest), Superior, Advanced, Intermediate, and Novice (lowest).
Change in Health Coach Interpersonal Communication from Baseline to 6 Months as Assessed by the RIAS | From baseline to 6 months
  Numerical score measured by the Roter Interaction Analysis System (RIAS).

OTHER OUTCOMES:
Change in Program Acceptability from Baseline to End of Year 5 | From baseline to end of Year 5
  Qualitative interviews with academic faculty reported as qualitative themes.
Change in Program Reach to End of Year 5 | From baseline to end of Year 5
  Number of students by academic program reported as numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Usha Menon, PhD, RN,, Principal Investigator — University of South Florida College of Nursing; Glenn A Martinez, PhD, MPH, Principal Investigator — The University of Texas at San Antonio
Locations (2):
- United States (2):
  - University of Arizona College of Nursing, Tucson, Arizona
  - The Ohio State University College of Arts and Sciences, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified data obtained through this study will be available upon request to share with qualified students and faculty engaging in independent scientific research.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to four years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to de-identified Individual Participant Data from this trial can be requested if the requestor obtains the appropriate clearance from their Institutional Review Board for the secondary analysis project and if the requestor is willing to complete a Data Sharing Agreement. For more information or to submit a request, please contact Dr. Usha Menon at umenon@usf.edu.

REFERENCES:
- [Result] Menon U, Szalacha LA, Martinez GA, Graham MC, Pares-Avila JA, Rechenberg K, Stauber LS. Efficacy of a language-concordant health coaching intervention for latinx with diabetes. Patient Educ Couns. 2022 Jul;105(7):2174-2182. doi: 10.1016/j.pec.2021.11.024. Epub 2021 Nov 28. PMID 34895775